CLINICAL TRIAL: NCT06959550
Title: Phase II Study of Anti-PD-1/VEGF Bispecific Antibody Ivonescimab in Patients With Previously Treated Metastatic Colorectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Akesobio Australia Pty Ltd (Industry); Summit Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0278; NCI-2025-03211 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2025-04-28; First posted 2025-05-06 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment with Ivonescimab (Experimental): Participants will be assigned to the study using a Bayesian Optimal Phase 2 (BOP2) design
  Interventions: Drug: Ivonescimab

INTERVENTIONS:
Drug: Ivonescimab — Given by IV

SUMMARY:
The goal of this clinical research study is to learn if ivonescimab can help to control previously treated, metastatic colorectal cancer.

DETAILED DESCRIPTION:
Primary Objective:

• To evaluate the efficacy of ivonescimab, as determined by the objective response rate per iRECIST, in three distinct cohorts of patients with treatment-refractory metastatic colorectal cancer: 1) dMMR/MSI-H refractory to anti-PD-1 therapy, 2) pMMR/MSS without liver metastases, and 3) pMMR/MSS with liver metastases.

Secondary Objective:

* To evaluate the safety of ivonescimab in patients with metastatic colorectal cancer.
* To evaluate the efficacy of ivonescimab, as determined by the objective response rate per RECIST 1.1, in three distinct cohorts of patients with treatment-refractory metastatic colorectal cancer: 1) dMMR/MSI-H refractory to anti-PD-1 therapy, 2) pMMR/non-MSI-H without liver metastases, and 3) pMMR/non-MSI-H with liver metastases.
* To evaluate changes in intratumoral CD8+ T cell density following ivonescimab therapy.

Exploratory Objectives:

* To assess the time to response following treatment with ivonescimab in patients with metastatic colorectal cancer.
* To assess the durability of response following treatment with ivonescimab in patients with metastatic colorectal cancer.
* To evaluate progression-free survival following treatment with ivonescimab in patients with metastatic colorectal cancer.
* To evaluate overall survival following treatment with ivonescimab in patients with metastatic colorectal cancer.
* To investigate clinical, pathologic, and molecular features associated with therapeutic response to ivonescimab in patients with metastatic colorectal cancer.
* To investigate changes in immune cell composition and distance relationships within the metastatic CRC tumor microenvironment following ivonescimab therapy.
* To evaluate changes in peripheral immune cell populations in metastatic CRC patients following ivonescimab therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving signed informed consent
2. Male and female adult participants 18 years of age or older on day of signing informed consent.
3. Histological or cytological confirmed advanced, metastatic adenocarcinoma of colon or rectum.
4. Known MMR or MSI status performed by local standard of practice. (e.g., IHC and/or PCR, next-generation sequencing)
5. Cohort-specific criteria

   * Cohort 1: MSI-H/dMMR: ICI-refractory

     * dMMR or MSI-H per local testing
     * Demonstrated radiographic or clinical disease progression following treatment with immune checkpoint inhibitors including anti-PD-1 +/- anti-CTLA-4 therapy. If progression occurred after first imaging assessment, then pseudo-progression should be excluded by concurrent carcinoembryonic antigen (CEA) or other tumor marker or ctDNA elevation, or clinical symptom progression, or short-interval repeat imaging confirming progression.
     * Must have received at least 2 doses of a PD1/PD-L1 inhibitor.
     * Progressive disease either during therapy or within 3 months of last dose of therapy.
     * No serious adverse immune-related adverse events (grade 3 or higher) with previous immune checkpoint therapy, that were symptomatic and required prolonged immunosuppression (>6 weeks).
   * Cohort 2: pMMR with liver metastases

     * pMMR or non-MSI-H per local testing
     * Presence of active liver metastases per radiographic imaging
     * Patients with any bulky liver metastases measuring >5.0 cm are not eligible
   * Cohort 3: pMMR without liver metastases

     * pMMR or non-MSI-H per local testing
     * No liver metastases per radiographic imaging (note: previously treated or resected liver metastases are allowed if treatment was >6 months prior without liver progression)
6. Known extended RAS and BRAF status as per local standard of practice (Cohorts 2 and 3 only)
7. Participant must have progressed (radiologically or clinically) or been intolerant to fluoropyrimidine, irinotecan, and oxaliplatin (Cohorts 2 and 3 only)

   * Patient must have evidence of progression on or after the last treatment regimen received and within 6 months prior to study enrollment
   * Patients who were intolerant to prior systemic chemotherapy regimens are eligible if there is documented evidence of clinically significant intolerance despite adequate supportive measures.
   * Perioperative chemotherapy exposure can be considered if the participant had disease recurrence within 12 months of completion of neoadjuvant chemotherapy or 6 months of completion of adjuvant chemotherapy
8. ECOG (Eastern Cooperative Oncology Group) PS of 0 to 1.
9. Adequate hematologic and organ function as assessed by the following laboratory tests performed within 7 days before treatment initiation:

   * Total bilirubin .1.5 x the upper limit of normal (ULN). Total bilirubin (.3 x ULN) is allowed if Gilbert fs syndrome is documented.
   * Alanine transaminase (ALT) and aspartate aminotransferase (AST) .2.5x ULN (.5 x ULN for patients with liver involvement of their cancer)
   * Platelet count .100,000 /mm3, Hemoglobin (Hb) .9 g/dL, WBC .2000/ƒÊL absolute neutrophil count (ANC) .1500/mm3 without red blood cell transfusion or growth factor administered within 7 days of screening CBC.
   * Serum creatinine .1.5 x ULN or creatinine clearance .50 mL/min (measured or calculated using the Cockroft-Gault formula)
   * Prothrombin time-international normalized ratio (PT/INR) . 1.5 x ULN and partial prothrombin time (PTT) or activated partial thromboplastin time (aPTT) . 1.5 ~ ULN (unless abnormalities are unrelated to coagulopathy) This applies only to patients who are not on therapeutic anti-coagulation. Patients receiving therapeutic anti-coagulation should be on a stable dose.
   * Estimated CrCl . 50 mL/min.
   * Proteinuria . 30 mg/dL.
10. Measurable disease as determined by iRECIST v1.1.
11. Ability to provide recent tumor tissue is mandatory for all participants at screening, either through pre-treatment biopsy or archived tissue. For archived tissue, FFPE block or a minimum of 10 slides is recommended with exceptions to these criteria permitted for consideration by the principal investigator.
12. Anticipated life expectancy greater than 3 months
13. Women of childbearing potential (WOCBP) must agree to follow instructions for method(s) of contraception for the duration of study intervention and 4 months after the last dose of study drug. Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of study intervention and 4 months after the last dose of study drug. In addition, male participants must be willing to refrain from sperm donation during this time. Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Exclusion Criteria:

1. Any single liver metastasis >5.0 cm (Cohort 2 only)
2. Except for MSI-H/dMMR tumors, prior therapy with PD-1, PD-L1, or CTLA-4 inhibitors (Cohorts 2 and 3 only).
3. Patient who discontinued prior therapy with immune checkpoint inhibitors due to Grade 2 neurologic, cardiac, or ophthalmologic events or recurrent Grade 2 pneumonitis are not eligible for the trial (Cohort 1 only).
4. Systemic anti-cancer treatment within 14 days or less than 5 half-lives (whichever is shorter) of the first dose of study treatment.
5. Has unresolved clinically significant toxicity of greater than or equal to NCI Institute Common Terminology Criteria for AEs (CTCAE v5.0) grade 2 attributed to any prior therapies (excluding anemia, lymphopenia, alopecia, skin pigmentation, and immune toxicities for MSI-H/dMMR ICI-refractory cohort as listed in cohort inclusion criteria).
6. History of arterial thromboembolic event, venous thromboembolic event of grade 3 and above as specified in NCI CTCAE v5.0, transient ischemic attack, cerebrovascular accident, hypertensive crisis, or hypertensive encephalopathy within 12 months prior to enrollment
7. Unstable angina, myocardial infarction, congestive heart failure (New York Heart Association [NYHA] classification . grade 2) or unstable vascular disease (eg, aortic aneurysm at risk of rupture, Moyamoya disease) that required hospitalization within 12 months prior to randomization, or other cardiac impairment that may affect the safety evaluation of the study drug (eg, poorly controlled arrhythmias, myocardial ischemia)
8. Acute exacerbation of chronic obstructive pulmonary disease within 4 weeks before enrollment
9. Poorly controlled hypertension with repeated systolic blood pressure . 150 mmHg or diastolic blood pressure . 100 mmHg after oral antihypertensive therapy
10. Active autoimmune or lung disease requiring systemic therapy (eg, with disease modifying drugs, prednisone >10 mg daily or equivalent, immunosuppressant therapy) within 2 years prior to randomization, however the following will be allowed: a. Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is permitted. b. Intermittent use of bronchodilators, inhaled corticosteroids, or local corticosteroid injections is permitted
11. Know history of esophageal gastric varices, severe ulcers, wounds that do not heal, abdominopelvic fistula, intra-abdominal abscesses, or acute gastrointestinal bleeding within 6 months prior to enrollment
12. History of perforation of the gastrointestinal tract and/or fistula, gastrointestinal obstruction (including incomplete intestinal obstruction requiring parenteral nutrition), or extensive bowel resection (partial colectomy or extensive small bowel resection) within 6 months prior to enrollment
13. History of bleeding tendencies or coagulopathy and/or clinically significant bleeding symptoms or risk within 4 weeks prior to enrollment, including but not limited to:

    * Hemoptysis (defined as coughing up . 0.5 teaspoon of fresh blood or small blood clots. Note: transient hemoptysis associated with diagnostic bronchoscopy is allowed
    * Nasal bleeding/epistaxis (bloody nasal discharge is allowed)
    * Current use of prophylactic or full-dose anticoagulants or anti-platelet agents for therapeutic purposes that is not stable prior to enrollment is not permitted. The use of full-dose anticoagulants is permitted if the international normalized ratio (INR) or activated partial thromboplastin time (aPTT) is within therapeutic limits according to the medical standard of the enrolling institution.
14. Subjects whose tumors invade peripheral important organs and blood vessels (such as heart and pericardium, trachea, esophagus, aorta, superior vena cava, etc), and who are at risk of esophageal tracheal fistula or esophageal pleural fistula or intestinal fistula
15. Symptomatic CNS metastases, CNS metastases with hemorrhagic features, CNS metastasis . 1.5 cm, CNS radiation within 7 days prior to randomization, potential need for CNS radiation within the first cycle, or leptomeningeal disease. Note: Patients must have stopped corticosteroids or be on physiologic corticosteroid replacement therapy (prednisone .10 mg daily or equivalent).
16. Live vaccine or live attenuated vaccine within 4 weeks prior to planned enrollment, or if scheduled to receive a live vaccine or live attenuated vaccine during the study period. Inactivated vaccines are permitted.
17. Severe infection within 4 weeks prior to enrollment, including but not limited to comorbidities requiring hospitalization, sepsis, or severe pneumonia; active infection (as determined by the investigator) requiring systemic anti-infective therapy within 2 weeks prior to enrollment. Participants with HIV, HCV, or HBV infection may be included if suppressive antiviral therapy has been administered and the viral load is undetectable.
18. Has pre-existing peripheral neuropathy that is . grade 2 per NCI CTCAE v5.0.
19. Major surgical procedures or serious trauma within 4 weeks prior to enrollment, or plans for major surgical procedures within 4 weeks after the first dose (as determined by the investigator). Minor local procedures (excluding central venous catheterization and port implantation) within 3 days prior to enrollment.
20. Uncontrolled pleural effusions, pericardial effusions, or ascites that is clinically symptomatic. Note: Patients managed with indwelling catheters (e.g. PleurX) are allowed.
21. History of non-infectious pneumonia requiring systemic corticosteroids, or current interstitial lung disease
22. Active or prior history of inflammatory bowel disease (eg, Crohn fs disease, ulcerative colitis, or chronic diarrhea)
23. Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation
24. Known allergy to any component of any study drug or known history of severe hypersensitivity to other monoclonal antibodies
25. Has any other clinically significant cardiac, respiratory, or other medical or psychiatric condition that might interfere with participation in the trial or interfere with the interpretation of trial results, in the opinion of the investigator.
26. Participants with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of start of study treatment. Inhaled or topical steroids, and adrenal replacement steroid doses >10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
27. Pregnancy or breast feeding.
28. Psychological, familial, or sociological condition potentially hampering compliance with the study protocol and follow-up schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-07-28 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2030-07-01 (Estimated)

PRIMARY OUTCOMES:
1. Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Saurav Haldar, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org